CLINICAL TRIAL: NCT00266227
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study of Retreatment With Rituximab in Subjects With Rheumatoid Arthritis Receiving Background Methotrexate
Brief Title: A Study of Retreatment With Rituximab in Patients With Rheumatoid Arthritis Receiving Background Methotrexate
Acronym: SUNRISE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: U3384g
Record Dates: First submitted 2005-12-14; First posted 2005-12-16 (Estimated); Results first posted 2009-05-25 (Estimated); Last update posted 2013-10-25 (Estimated); Status verified 2013-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Rituximab; Methotrexate; Folic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Arm A: Rituximab Retreatment (Experimental): 1000 mg rituximab intravenous initial treatment on day 1 and day 15 plus 10-25 mg/week methotrexate followed by re-treatment during weeks 24 -40 consisting of two additional doses of 1000 mg rituximab 14 days apart plus 10-25 mg/week methotrexate.
  Interventions: Drug: rituximab; Drug: methotrexate; Drug: folate
- Arm B: Placebo Retreatment (Placebo Comparator): 1000 mg rituximab intravenous initial treatment on day 1 and day 15 plus 10-25 mg/week methotrexate followed by retreatment during weeks 24 -40 consisting of two doses of placebo 14 days apart plus 10-25 mg/week methotrexate.
  Interventions: Drug: placebo; Drug: methotrexate; Drug: folate

INTERVENTIONS:
Drug: placebo — Intravenous repeating dose
  Arms: Arm B: Placebo Retreatment
Drug: rituximab — Intravenous repeating dose
  Arms: Arm A: Rituximab Retreatment
Drug: methotrexate — Oral or parenteral repeating dose
Drug: folate — Intravenous repeating dose

SUMMARY:
This is a Phase III, randomized, double-blind, placebo-controlled, multicenter study evaluating the efficacy of retreatment with rituximab in subjects with active rheumatoid arthritis (RA) who are receiving Methotrexate (MTX).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form
* Ability and willingness to comply with the requirements of the study protocol
* Age 18-80 years
* Diagnosis of RA for at least 6 months
* Receiving treatment for RA on an outpatient basis
* Documented moderate to severe active RA activity at screening and Day 1
* Documented inadequate response to previous or current treatment with one or more of the following: etanercept, infliximab, and/or adalimumab because of toxicity or inadequate efficacy
* Use of MTX 10-25 mg/wk for ≥ 12 weeks prior to Day 1 at a stable dose for ≥ 4 weeks
* Willingness to receive oral folic acid
* If taking a background corticosteroid, use of the corticosteroid must be at a stable dose during the 4 weeks prior to Day 1
* Use of one NSAID is permitted if the dose is stable for ≥ 2 weeks prior to Day 1
* For men and women of reproductive potential, willingness to use a reliable means of contraception for ≥ 30 days prior to Day 1 and for the study duration or the duration that the subject's peripheral CD19 B cells are depleted, whichever is longer

Exclusion Criteria:

* Rheumatic autoimmune disease other than RA or significant systemic involvement secondary to RA; Secondary Sjogren's syndrome with RA is permitted.
* History of or current inflammatory joint disease other than RA or other systemic rheumatic disorder (e.g., systemic lupus erythematosus, inflammatory bowel disease, scleroderma, inflammatory myopathy, or overlap syndrome)
* History of deep space/tissue infection within 52 weeks prior to Day 1
* Diagnosis of juvenile idiopathic arthritis (JIA), juvenile rheumatoid arthritis (JRA), and/or RA before age 16
* Functional Class IV, as defined by the ACR Classification of Functional Status in Rheumatoid Arthritis
* Any surgical procedure, including bone/joint surgery/synovectomy (including joint fusion or replacement), within 12 weeks prior to Day 1 or planned within 48 weeks after Day 1
* Known hypersensitivity to any component of a humanized or murine monoclonal antibody
* Receipt of any vaccination within 4 weeks prior to Day 1
* Significant cardiac or pulmonary disease, including obstructive pulmonary disease
* Evidence of significant uncontrolled concomitant disease, such as, but not limited to nervous system, renal, hepatic, endocrine, or gastrointestinal disorders
* Known active bacterial, viral, fungal, mycobacterial, or other infection (including tuberculosis or atypical mycobacterial disease but excluding fungal infections of the nail beds) or any major episode of infection requiring hospitalization or treatment with IV antibiotics within 4 weeks of Day 1 or oral antibiotics within 2 weeks of Day 1
* History of serious recurrent or chronic infection (a chest X-ray will be performed at screening if one has not been performed within 12 weeks of screening that showed no clinically significant abnormality)
* History of or currently active primary or secondary immunodeficiency, including HIV infection
* History of cancer, including solid tumors and hematologic malignancies (except basal cell or squamous cell carcinoma of the skin that has been excised and cured)
* History of significant cytopenias or other bone marrow disorders
* History of alcohol, drug, or chemical abuse within 24 weeks prior to Day 1
* Pregnancy or lactation
* Neuropathies and neurovasculopathies that might interfere with pain evaluation
* Poor peripheral venous access
* Intolerance or contraindications to oral or IV corticosteroids
* Positive hepatitis B surface antigen or hepatitis C antibody serology
* For women of childbearing potential (including those who have had a tubal ligation), a positive serum pregnancy test at screening
* Current use of any DMARD other than MTX
* Concurrent treatment with any biologic agent
* Treatment with any investigational agent within 4 weeks prior to Day 1 or five half-lives of the investigational drug (whichever is longer)
* Any previous treatment with rituximab or other cell-depleting therapies, including CAMPATH, anti-CD4, anti-CD5, anti-CD3, anti-CD19, anti-CD11a, anti-CD22, anti-BLys/ BAFF, and other anti-CD20 agents
* Previous treatment with a co-stimulation blocking agent, including abatacept
* Previous treatment with an anti-<alpha> 4 integrin agent, including natalizumab
* Previous treatment within 6 months of screening with IV & globulin or the Prosorba(R) Column
* Intra-articular or parenteral corticosteroids within 4 weeks prior to Day 1

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 559 (Actual)
Dates: Start 2006-01; Primary Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anshu Vashishtha, MD PhD, Study Director — Genentech, Inc.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 559 participants received initial treatment open label rituximab. 84 of these participants were not randomized to Retreatment.
Groups:
- Rituximab-Not Randomized to Retreatment: 1000 mg rituximab intravenous initial treatment on day 1 and day 15 plus 10-25 mg/week methotrexate. Participants were not randomized to Retreatment.
Period: Initial Treatment
Arm/Group | Arm A: Rituximab Retreatment | Arm B: Placebo Retreatment | Rituximab-Not Randomized to Retreatment
Started | 0 | 0 | 559
Completed | 0 | 0 | 482
Not Completed | 0 | 0 | 77
Not completed — Adverse Event | 0 | 0 | 13
Not completed — Lost to Follow-up | 0 | 0 | 6
Not completed — Subject/Guardian decision to withdraw | 0 | 0 | 45
Not completed — Physician decision to withdraw | 0 | 0 | 12
Not completed — Pregnancy | 0 | 0 | 1
Period: Retreatment: Up to Week 48
Arm/Group | Arm A: Rituximab Retreatment | Arm B: Placebo Retreatment | Rituximab-Not Randomized to Retreatment
Started | 318 | 157 | 0
Completed | 291 | 134 | 0
Not Completed | 27 | 23 | 0
Not completed — Death | 1 | 0 | 0
Not completed — Adverse Event | 7 | 7 | 0
Not completed — Lost to Follow-up | 3 | 0 | 0
Not completed — Subject/Guardian Decision to Withdraw | 11 | 14 | 0
Not completed — Physician's Decision to Withdraw | 4 | 2 | 0
Not completed — Pregnancy | 1 | 0 | 0
Period: Retreatment: Week 48 to Week 72
Arm/Group | Arm A: Rituximab Retreatment | Arm B: Placebo Retreatment | Rituximab-Not Randomized to Retreatment
Started | 291 | 134 | 0
Completed | 227 | 92 | 0
Not Completed | 64 | 42 | 0
Not completed — Death | 1 | 1 | 0
Not completed — Adverse Event | 6 | 2 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Subject/Guardian Decision to Withdraw | 41 | 29 | 0
Not completed — Physician's Decision to Withdraw | 15 | 10 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm B: Placebo Retreatment: 1000 mg rituximab initial treatment on day 1 and day 15 plus 10-25 mg/wk methotrexate followed by re-treatment during weeks 24 -40 consisting of two doses of placebo 14 days apart plus 10-25 mg/wk methotrexate.
- Total: Total of all reporting groups
Arm/Group | Arm A: Rituximab Retreatment | Arm B: Placebo Retreatment | Total
Number analyzed (Participants) | 318 | 157 | 475
Age, Categorical [Count of Participants; unit: Participants] — Baseline measures are based on the Intent-to-treat population that includes all participants randomized to Retreatment.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 266 | 133 | 399
    >=65 years | 52 | 24 | 76
Age Continuous [Mean (Standard Deviation); unit: years] | 54.2 (10.57) | 53.9 (10.52) | 54.1 (10.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 257 | 124 | 381
  Male | 61 | 33 | 94

OUTCOME MEASURES:

1. Primary Outcome: Retreated Subjects With an American College of Rheumatology 20% (ACR20) Response at Week 48 Relative to Baseline
Description: ACR20 response was defined as a ≥ 20% improvement compared with baseline in both tender joint count (TJC) [68 joints] and swollen joint count (SJC) [66 joints] as well as a ≥ 20% improvement in three of five additional measurements: 1) Physician's Global Assessment of disease activity [visual analog scale: 0=no disease activity to 100=maximum disease activity]; 2) Patient's Global Assessment of Disease Activity [visual analog scale: 0=no disease activity to 100=maximum disease activity]; 3) Patient's Assessment of Pain [visual analog scale: 0=no pain to 100=unbearable pain]; 4) Health Assessment Questionnaire [20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities, 0=without difficulty to 3=unable to do] and 5) erythrocyte sedimentation rate.
Time Frame: 48 Weeks
Population: Intent-to-treat population includes all participants randomized to Retreatment.
Measure: Number; unit: Participants
Arm/Group | Arm A: Rituximab Retreatment | Arm B: Placebo Retreatment
Number analyzed (Participants) | 318 | 157
Participants | 170 [48.0 to 58.9] | 70
Statistical Analysis 1: Comparison: Arm A: Rituximab Retreatment vs Arm B: Placebo Retreatment; Test type: Superiority or Other; p = 0.0195, Cochran-Mantel-Haenszel

2. Secondary Outcome: Retreated Subjects With American College of Rheumatology 50% (ACR50) Response and American College of Rheumatology 70% (ACR70) Response at Week 48 Relative to Baseline
Description: ACR50 or ACR70 response was defined as a ≥ 50% or 70% improvement compared with baseline in both tender joint count (TJC) [68 joints] and swollen joint count (SJC) [66 joints] as well as a ≥ 50% or 70% improvement in three of five additional measurements: 1) Physician's Global Assessment of disease activity [visual analog scale: 0=no disease activity to 100=maximum disease activity]; 2) Patient's Global Assessment of Disease Activity [visual analog scale: 0=no disease activity to 100=maximum disease activity]; 3) Patient's Assessment of Pain [visual analog scale: 0=no pain to 100=unbearable pain]; 4) Health Assessment Questionnaire [20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities, 0=without difficulty to 3=unable to do] and 5) erythrocyte sedimentation rate.
Time Frame: Baseline, Week 48
Population: Intent-to-treat population includes all participants randomized to Retreatment.
Measure: Number; unit: Participants
Arm/Group | Arm A: Rituximab Retreatment | Arm B: Placebo Retreatment
Number analyzed (Participants) | 318 | 157
Participants
  ACR50 | 92 [23.9 to 33.9] | 41
  ACR70 | 44 [10.0 to 17.6] | 21

3. Secondary Outcome: Change From Baseline in the Disease Activity Score Using 28 Joint Counts (DAS28-ESR) at Week 48
Description: The DAS28 score is a measure of the patient's disease activity calculated using the tender joint count (TJC) [28 joints], swollen joint count (SJC) [28 joints], patient's global assessment of disease activity [visual analog scale: 0=no disease activity to 100=maximum disease activity] and the erythrocyte sedimentation rate (ESR) for a total possible score of 2 to 10. Higher values indicate higher disease activity. A negative change from baseline indicates improvement.
Time Frame: 48 weeks
Population: Participants from the Intent-to-treat population, that includes all participants randomized to Retreatment, with data available for analyses.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Arm A: Rituximab Retreatment | Arm B: Placebo Retreatment
Number analyzed (Participants) | 312 | 157
Units on a scale | -2.1 (1.55) | -1.8 (1.69)
Statistical Analysis 1: Comparison: Arm A: Rituximab Retreatment vs Arm B: Placebo Retreatment; Assessed using an analysis of variance (ANOVA) model, with retreatment group, baseline DAS28-ESR score, baseline RF status, and ≥20% improvement in both SJC and TJC at Week 24 from baseline (yes/no) as explanatory terms in the model; Test type: Superiority or Other; ANOVA; Adjusted mean for Arm A (Rituxan) is -1.9 and adjusted mean for Arm B (Placebo) is -1.5; Mean Difference (Final Values) = -0.4, 95% CI [-0.7 to -0.1]

4. Secondary Outcome: Change From Baseline in Disease Activity Score (DAS28-CRP) at Week 48
Description: The DAS28 score is a measure of the patient's disease activity calculated using the tender joint count (TJC) [28 joints], swollen joint count (SJC) [28 joints], patient's global assessment of disease activity [visual analog scale: 0=no disease activity to 100=maximum disease activity] and C-Reactive Protein (CRP) for a total possible score of 2 to 10. Higher values indicate higher disease activity. A negative change from baseline indicates improvement.
Time Frame: Baseline, Week 48
Population: Participants from the Intent-to-treat population that includes all participants randomized to Retreatment with data available for analyses.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Arm A: Rituximab Re-treatment: 1000 mg rituximab intravenous initial treatment on day 1 and day 15 plus 10-25 mg/week methotrexate followed by re-treatment during weeks 24 -40 consisting of two additional doses of 1000 mg rituximab 14 days apart plus 10-25 mg/week methotrexate.
- Arm B: Placebo Re-treatment: 1000 mg rituximab initial treatment on day 1 and day 15 plus 10-25 mg/wk methotrexate followed by re-treatment during weeks 24 -40 consisting of two doses of placebo 14 days apart plus 10-25 mg/wk methotrexate.
Arm/Group | Arm A: Rituximab Re-treatment | Arm B: Placebo Re-treatment
Number analyzed (Participants) | 316 | 157
Units on a scale | -1.8 (1.4) | -1.5 (1.5)

5. Secondary Outcome: Percentage of Retreated Subjects With a European League Against Rheumatism (EULAR) Response at Week 48
Description: Change of the Disease Activity Score 28 score from baseline was used to determine EULAR responses of good, moderate, or no response. For a post-baseline score ≤ 3.2, a change from baseline of < -1.2 was a good response, < -0.6 to ≥ -1.2 was a moderate response, and ≥ -0.6 was no response. For a post-baseline score > 3.2 to ≤ 5.1, a change from baseline of < -0.6 was a moderate response and ≥ -0.6 was no response. For a post-baseline score > 5.1, a change from baseline < -1.2 was a moderate response and ≥ -1.2 was no response. A good response could not be achieved for post-baseline scores > 3.2.
Time Frame: Baseline, Week 48
Population: Intent-to-treat population includes all participants randomized to Retreatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Arm A: Rituximab Retreatment | Arm B: Placebo Retreatment
Number analyzed (Participants) | 318 | 157
Percentage of participants
  Good Response | 20.8 | 18.5
  Moderate Response | 47.5 | 42.7

6. Secondary Outcome: Change From Baseline in American College of Rheumatology (ACR) Core Set Component: Swollen Joint Count at Week 48
Description: A Rheumatologist or an skilled arthritis assessor evaluated 66 joints at baseline and at Week 48. A negative change from baseline in Swollen Joint Count indicates improvement.
Time Frame: Baseline, Week 48
Population: Intent-to-treat population includes all participants randomized to Retreatment.
Measure: Mean (Standard Deviation); unit: Joint Count
Arm/Group | Arm A: Rituximab Retreatment | Arm B: Placebo Retreatment
Number analyzed (Participants) | 318 | 157
Joint Count | -12.5 (12.31) | -10.2 (13.30)

7. Secondary Outcome: Change From Baseline in American College of Rheumatology (ACR) Core Set Component: Tender Joint Count at Week 48
Description: A Rheumatologist or an skilled arthritis assessor evaluated 68 joints at baseline and at Week 48. A negative change from baseline in the Tender Joint Count indicates improvement.
Time Frame: Baseline, Week 48
Population: Intent-to-treat population includes all participants randomized to Retreatment.
Measure: Mean (Standard Deviation); unit: Joint Count
Arm/Group | Arm A: Rituximab Retreatment | Arm B: Placebo Retreatment
Number analyzed (Participants) | 318 | 157
Joint Count | -15.3 (15.28) | -14.7 (18.71)

8. Secondary Outcome: Change From Baseline in American College of Rheumatology (ACR) Core Set Component: Health Assessment Questionnaire Disability Index (HAQ-DI) at Week 48
Description: The Stanford Health Assessment Questionnaire disability index (HAQ-DI) is a patient completed questionnaire specific for rheumatoid arthritis. It consists of 20 questions referring to 8 domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip,and common daily activities. Each domain has at least two component questions. There are four possible responses for each component ranging from 0(without any difficulty) to 4 (unable to do).HAQ-DI=sum of worst scores in each domain divided by the number of domains answered. A negative change from baseline indicates improvement.
Time Frame: Baseline, Week 48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Arm A: Rituximab Retreatment | Arm B: Placebo Retreatment
Number analyzed (Participants) | 316 | 157
Score on a scale | -0.3 (0.53) | -0.2 (0.60)

9. Secondary Outcome: Change From Baseline in American College of Rheumatology (ACR) Core Set Component: Subject's Global Assessment of Disease Activity at Week 48
Description: Participants rated their disease activity at baseline and Week 48 using the Visual Analog Scale (VAS) on a scale of 0 (best) to 100 (worse). A negative change from baseline indicates improvement.
Time Frame: Baseline, Week 48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: millimeter (mm)
Arm/Group | Arm A: Rituximab Retreatment | Arm B: Placebo Retreatment
Number analyzed (Participants) | 316 | 157
millimeter (mm) | -26.9 (29.04) | -23.0 (28.72)

10. Secondary Outcome: Change From Baseline in American College of Rheumatology (ACR) Core Set Component: Physician's Global Assessment of Disease Activity at Week 48
Description: A Rheumatologist or a skilled Arthritis assessor rated the patient's disease activity at baseline and Week 48 using the Visual Analog Scale (VAS) on a scale of 0 (best) to 100 (worse). A negative change from baseline indicates improvement.
Time Frame: Baseline, Week 48
Population: Intent-to-treat population includes all participants randomized to Retreatment.
Measure: Mean (Standard Deviation); unit: millimeter (mm)
Arm/Group | Arm A: Rituximab Retreatment | Arm B: Placebo Retreatment
Number analyzed (Participants) | 318 | 157
millimeter (mm) | -31.5 (27.00) | -25.5 (29.59)

11. Secondary Outcome: Change From Baseline in American College of Rheumatology (ACR) Core Set Component: Subject's Assessment of Pain at Week 48
Description: Patients rated their pain at baseline and Week 48 using the Visual Analog Scale (VAS) on a scale of 0 (none) to 100 (unbearable pain). A negative change from baseline indicates improvement.
Time Frame: Baseline, Week 48
Population: Participants from the Intent-to-treat population, that includes all participants randomized to Retreatment with data available for analyses.
Measure: Mean (Standard Deviation); unit: millimeter (mm)
Arm/Group | Arm A: Rituximab Retreatment | Arm B: Placebo Retreatment
Number analyzed (Participants) | 317 | 157
millimeter (mm) | -24.0 (28.99) | -19.3 (30.32)

12. Secondary Outcome: Change From Baseline in American College of Rheumatology (ACR) Core Set Component: C-Reactive Protein at Week 48
Description: Blood was collected for C-Reactive Protein, an inflammatory marker, at Baseline and Week 48. A negative change from baseline indicates improvement.
Time Frame: Baseline, Week 48
Population: Intent-to-treat Population includes all participants randomized to Retreatment.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Arm A: Rituximab Retreatment | Arm B: Placebo Retreatment
Number analyzed (Participants) | 318 | 157
mg/dL | -0.8 (2.55) | -0.6 (2.95)

13. Secondary Outcome: Change From Baseline in American College of Rheumatology (ACR) Core Set Component: Erythrocyte Sedimentation (ESR) at Week 48
Description: Blood was collected for Erythrocyte Sedimentation Rate, an inflammatory marker, at Baseline and Week 48. A negative change from baseline indicates improvement.
Time Frame: Baseline, Week 48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: millimeter/hour (mm/hr)
Arm/Group | Arm A: Rituximab Retreatment | Arm B: Placebo Retreatment
Number analyzed (Participants) | 315 | 157
millimeter/hour (mm/hr) | -15.0 (25.03) | -10.9 (24.00)

14. Secondary Outcome: Percentage of Retreated Subjects With a Change ≥ 0.22 From Baseline in HAQ-DI at Week 48
Description: The Stanford Health Assessment Questionnaire disability index (HAQ-DI) is a patient completed questionnaire specific for rheumatoid arthritis. It consists of 20 questions referring to 8 domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip and common daily activities. Each domain has at least two component questions. There are four possible responses for each component ranging from 0(without any difficulty) to 4 (unable to do). HAQ-DI=sum of worst scores in each domain divided by the number of domains answered.
Time Frame: Baseline, Week 48
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Arm A: Rituximab Re-treatment | Arm B: Placebo Re-treatment
Number analyzed (Participants) | 316 | 157
Percentage of participants | 57.3 | 51.0

15. Secondary Outcome: Percentage of Retreated Subjects With a Change ≥ 0.3 From Baseline in HAQ-DI at Week 48
Description: The Stanford Health Assessment Questionnaire disability index (HAQ-DI) is a patient completed questionnaire specific for rheumatoid arthritis. It consists of 20 questions referring to 8 domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip and common daily activities. Each domain has at least two component questions. There are four possible responses for each component ranging from 0(without any difficulty) to 4 (unable to do).HAQ-DI=sum of worst scores in each domain divided by the number of domains answered.
Time Frame: Baseline, Week 48
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Arm A: Rituximab Re-treatment | Arm B: Placebo Re-treatment
Number analyzed (Participants) | 316 | 157
Percentage of participants | 45.9 | 39.5

16. Secondary Outcome: ACRn in Retreated Subjects at Week 48
Description: The ACRn is calculated for each participant by taking the lowest percentage improvement in (1) swollen joint count or (2) tender joint count or (3) the median of the remaining 5 components of the ACR response (participant's assessment of disease activity; participant's global assessment of pain; physician's assessment of disease activity; participant's assessment of physical function; an acute phase reactant value - CRP). A positive ACRn Score indicates an improvement.
Time Frame: Baseline, Week 48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Arm A: Rituximab Re-treatment | Arm B: Placebo Re-treatment
Number analyzed (Participants) | 317 | 157
Score on a scale | 22.1 (45.29) | 10.7 (62.08)

17. Secondary Outcome: Change From Baseline in SF-36 Health Summary Scores at Week 48 in Retreated Subjects
Description: The SF-36 is a questionnaire used to assess physical functioning and is made up of eight domains: Physical Functioning, Role Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role-Emotional and Mental Health. Transforming and standardizing these domains leads to the calculation of the Physical (PCS) and Mental (MCS) Component Summary measures. Scores ranging from 0 to 100, with 0=worst score (or quality of life) and 100=best score. A positive change from baseline indicates improvement.
Time Frame: Baseline, Week 48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Arm A: Rituximab Re-treatment | Arm B: Placebo Re-treatment
Number analyzed (Participants) | 312 | 154
Score on a scale
  Mental Health Score | 4.6 (11.80) | 3.9 (13.50)
  Physical Health Score | 6.4 (8.76) | 4.8 (8.97)

18. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy Fatigue (FACIT-F) at Week 48 in Retreated Subjects
Description: FACIT-F is a 13-item questionnaire. Patients scored each item on a 5-point scale: 0 (Not at all) to 4 (Very much). The larger the patient's response to the questions (with the exception of 2 negatively stated), the greater the patient's fatigue. For all questions, except for the 2 negatively stated ones, the code was reversed and a new score was calculated as (4 minus the patient's response). The sum of all responses resulted in the FACIT-Fatigue score for a total possible score of 0 (worse score) to 52 (better score). A higher score reflects an improvement in the patient's health status.
Time Frame: Baseline, Week 48
Population: Participants from the Intent-to-treat population, that includes all randomized participants, with data available for analyses.
Measure: Median (Full Range); unit: Score on a scale
Arm/Group | Arm A: Rituximab Re-treatment | Arm B: Placebo Re-treatment
Number analyzed (Participants) | 317 | 157
Score on a scale | -5.0 [-29.0 to 27.0] | -4.0 [-32.0 to 22.0]

19. Secondary Outcome: Percentage of Retreated Subjects Achieving DAS28-ESR Remission at Week 48
Description: DAS28-ESR remission was defined as a DAS28-ESR < 2.6
Time Frame: Week 48
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Arm A: Rituximab Re-treatment | Arm B: Placebo Re-treatment
Number analyzed (Participants) | 317 | 157
Percentage of participants | 10.4 | 8.9

20. Secondary Outcome: Percentage of Retreated Subjects Achieving DAS28-ESR Low Disease at Week 48
Description: The DAS28-ESR score is a measure of the subject's disease activity. It is based on the tender joint count (28 joints), swollen joint count (28 joints), patient's global assessment of disease activity (mm), and ESR. DAS28-ESR scores range from 0 - 10. Low disease activity is defined as achieving a DAS28-ESR score of less than or equal to 3.2.
Time Frame: Week 48
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Arm A: Rituximab Re-treatment | Arm B: Placebo Re-treatment
Number analyzed (Participants) | 317 | 157
Percentage of participants | 21.1 | 18.5

ADVERSE EVENTS:
Arm/Group | Arm A: Rituximab Retreatment | Arm B: Placebo Retreatment | Rituximab-Not Randomized to Retreatment
Serious Adverse Events (participants affected / at risk) | 42/320 | 19/155 | 9/84
Other Adverse Events (participants affected / at risk) | 291/320 | 148/155 | 71/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Rituximab Retreatment (N=320) | Arm B: Placebo Retreatment (N=155) | Rituximab-Not Randomized to Retreatment (N=84)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 2 | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0
Coronary artery occlusion (Cardiac disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0
Pericarditis (Cardiac disorders) | 1 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0 | 0
Oesophagitis ulcerative (Gastrointestinal disorders) | 1 | 0 | 0
Chest pain (General disorders) | 1 | 1 | 0
Death (General disorders) | 1 | 0 | 0
Hernia obstructive (General disorders) | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0
Biliary dyskinesia (Hepatobiliary disorders) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 6 | 1 | 0
Abdominal abscess (Infections and infestations) | 0 | 1 | 0
Abdominal wall abscess (Infections and infestations) | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Perirectal abscess (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 2 | 1 | 1
Arthritis bacterial (Infections and infestations) | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 1 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0
Human ehrlichiosis (Infections and infestations) | 1 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0
Device failure (Injury, poisoning and procedural complications) | 0 | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Rheumatiod arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Joint destruction (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Cauda equina syndrome (Nervous system disorders) | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
Rectocele (Reproductive system and breast disorders) | 1 | 0 | 0
Uterine prolapse (Reproductive system and breast disorders) | 0 | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 2 | 0
Iliac artery occlusion (Vascular disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Rituximab Retreatment (N=320) | Arm B: Placebo Retreatment (N=155) | Rituximab-Not Randomized to Retreatment (N=84)
Nausea (Gastrointestinal disorders) | 35 | 15 | 5
Diarrhoea (Gastrointestinal disorders) | 25 | 9 | 8
Fatigue (General disorders) | 33 | 9 | 8
Pyrexia (General disorders) | 21 | 4 | 4
Upper respiratory tract infection (Infections and infestations) | 71 | 32 | 8
Sinusitis (Infections and infestations) | 45 | 16 | 5
Nasopharyngitis (Infections and infestations) | 20 | 11 | 4
Urinary tract infection (Infections and infestations) | 44 | 17 | 6
Bronchitis (Infections and infestations) | 22 | 16 | 4
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 74 | 59 | 19
Back pain (Musculoskeletal and connective tissue disorders) | 27 | 11 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 27 | 21 | 7
Headache (Nervous system disorders) | 51 | 18 | 13
Dizziness (Nervous system disorders) | 26 | 2 | 2
Insomnia (Psychiatric disorders) | 20 | 9 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 22 | 14 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 22 | 15 | 10
Rash (Skin and subcutaneous tissue disorders) | 21 | 10 | 4
Flushing (Vascular disorders) | 22 | 2 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other